CLINICAL TRIAL: NCT03415594
Title: A Once-weekly, Repeated Dose, Placebo Controlled, Double Blind, Randomised Cross-over Trial Investigating Safety, Efficacy and Pharmacodynamics of FE 203799 in Patients With Short Bowel Syndrome With Intestinal Failure Requiring Parenteral Support Followed by an Additional Treatment Period in an Open Label Regimen.
Brief Title: Safety, Efficacy, PD of FE203799 in Short Bowel Syndrome on Parenteral Support
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlyPharma Therapeutics (Industry)
Collaborators: VectivBio AG (Industry)
Responsible Party: Sponsor
Organization: VectivBio AG (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GLY-311-2017
Record Dates: First submitted 2017-11-16; First posted 2018-01-30 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2020-02

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FE203799 5 mg (Experimental): FE203799 GLP-2 analogue, once weekly, subcutaneous administration
  Interventions: Drug: FE203799 GLP-2 analogue
- Placebo (Placebo Comparator): Placebo FE203799 GLP-2 analogue, once weekly, subcutaneous administration
  Interventions: Drug: FE203799 Placebo GLP-2 analogue
- FE203799 10 mg (Other): FE203799 GLP-2 analogue, once weekly, subcutaneous administration
  Interventions: Drug: FE203799 GLP-2 analogue

INTERVENTIONS:
Drug: FE203799 GLP-2 analogue — FE203799 5 mg subQ once weekly
  Arms: FE203799 5 mg
Drug: FE203799 Placebo GLP-2 analogue — Placebo subQ once weekly
  Arms: Placebo
Drug: FE203799 GLP-2 analogue — FE203799 10 mg subQ once weekly
  Arms: FE203799 10 mg

SUMMARY:
Part A:once weekly dosing for 4 weeks in patients with short bowel syndrome who require total parenteral nutrition; patients will complete period 1 and after a 6-10 week wash-out, they will enter period 2 (active treatment and placebo); Part B: treatment period 3, is an open label extension to part A and starts after a washout of 6-10 weeks after the last dose in treatment period 2. patients are dosed once weekly for 4 weeks.

DETAILED DESCRIPTION:
This trial is divided into 2 parts. Part A of this trial is a repeated dose, placebo controlled, double blind, randomised cross-over trial investigating safety, efficacy and PD of FE 203799 in 8-10 patients with SBS. Additionally, the plasma concentration of FE 203799 will be assessed for determination of the trough and post-dose concentration in SBS patients. The patients will receive a subcutaneous (SC) dose of 5 mg FE 203799 or placebo once weekly for 4 consecutive weeks, and after a washout period of 6-10 weeks, the alternate treatment will be administered once weekly for 4 consecutive weeks. Safety follow-up assessments will be performed 6-10 weeks after the last dose in each treatment period.

Part B of this trial, treatment period 3, is an open label extension to part A that will test a new dose. Following a washout period of 6-10 weeks after the last dose in treatment period 2, the new dose will be administered once weekly for 4 weeks. Safety follow-up assessments will be performed 4-6 weeks after the last dose in treatment period 3.

The first two administrations of trial drug in each treatment period will be performed at the clinic, while the third and fourth dose can be either self-administered by the patient or administered at the clinic if the patient prefers to travel to the site or other considerations make a site visit preferable.

Prior to each administration of trial drug, liver function parameters will be analysed and assessed. During each treatment period, patients who develop extremely high or persistently elevated liver enzymes following trial drug administration will be discontinued from the trial.

The patients will complete a diary during each treatment period with daily data on parenteral support (PS) usage, oral liquid intake at specific periods, trial drug administrations performed at home, local tolerability and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria

1. Males and females with SBS secondary to surgical resection of small intestine
2. 18-80 years of age
3. Body Mass Index (BMI) between 16.0 and 32.0
4. Patients with a jejuno- or ileostomy and a faecal wet weight excretion of at least 1500 g/day, as recorded within the last 18 months according to the patient's medical record
5. Parenteral support ≥3 times/week for ≥12 months according to the patient's medical record
6. At least 6 months since last surgical bowel resection
7. Willing to adhere to a defined oral intake of fluids on certain days as required by the protocol (and based on the individual's routine daily consumption)
8. Women of childbearing potential must agree to use an adequate method of contraception during the trial and for 60 days after the end-of-trial visit. Adequate methods of contraception include intrauterine device or hormonal contraception (oral contraceptive pill, depot injections or implant, transdermal depot patch or vaginal ring). To be considered sterilised or infertile, females must have undergone surgical sterilisation (bilateral tubectomy, hysterectomy or bilateral ovariectomy) or be post-menopausal (defined as at least 12 months amenorrhoea and confirmed with follicle-stimulating hormone [FSH] test)

Exclusion Criteria

1. Pregnancy or lactation
2. Positive results on the human immunodeficiency virus (HIV), hepatitis B and/or C tests
3. A history of clinically significant intestinal adhesions and/or chronic abdominal pain
4. Require chronic systemic narcotics for treatment of pain that exceeds an amount corresponding to 80 mg of morphine per day
5. History of cancer or clinically significant lymphoproliferative disease within ≤5 years, except for adequately treated basal cell skin cancer
6. History of gallstone within the past 3 years. Gallstones with subsequent cholecystectomy to resolve the issues is acceptable
7. Inflammatory bowel disease (IBD) patients who have NOT been on a stable drug treatment regimen for at least the past 4 weeks
8. Evidence of active IBD in the past 12 weeks
9. Visible blood in the stool within the last 3 months
10. Catheter sepsis experienced within the last 3 months
11. Decompensated heart failure (New York Heart Association [NYHA] class III-IV) and/or known coronary heart disease defined as unstable angina pectoris and/or myocardial infarction within the last 6 months prior to screening
12. Radiation enteritis, scleroderma or other condition of intestinal dysmotility, coeliac disease, refractory or tropical sprue
13. History of alcohol and/or drug abuse within the last 12 months
14. Inadequate hepatic function as defined by: bilirubin >upper limit of normal (ULN), alanine transaminase (ALT) or aspartate transaminase (AST) >2.0 × ULN; alkaline phosphatase (ALP) >2.5 × ULN; or international normalised ratio (INR) >1.5 × ULN
15. Inadequate renal function as defined by serum creatinine or blood urea nitrogen >2.5 × ULN
16. Unplanned hospitalisation of >24 hours duration within 1 month before the screening visit
17. Systemic corticosteroids, methotrexate, cyclosporine, tacrolimus, sirolimus, infliximab or other biologic therapy/immune modifiers within 30 days of screening
18. Any use of growth hormone, glutamine or growth factors such as native glucagon-like peptide 2 (GLP 2) or GLP 2 analogue within the last 3 months
19. Any use of antibiotics within the last 30 days
20. Participation in another clinical trial within the last 3 months and during this trial
21. Previously been randomised in this trial
22. Loss of blood or donation of blood or plasma >500 mL within 3 months prior to screening
23. Patient not capable of understanding or not willing to adhere to the trial visit schedules and other protocol requirements
24. For any other reason judged not eligible by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day -28 to Day 29
  Adverse events (AEs) as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Assessment of intestinal failure and gut absorption | Day -3 - Day 28
  Measurement of urinary output (ml)
Assessment of intestinal failure and gut absorption | Day -3 - Day 28
  Measurement of urinary sodium (mmol/d)
Assessment of intestinal failure and gut absorption | Day -3 - Day 29
  Measurement of Parenteral Support (L)
Assessment of intestinal failure and gut absorption | Day -3 - Day 28
  Measurement of oral fluids intake (L)
Assessment of intestinal failure and gut absorption | Day -3 and Day 29
  Changes from baseline in lean body mass by DEXA scan
Assessment of intestinal failure and gut absorption | Day -3 and Day 29
  Changes from baseline in fat mass by DEXA scan
Assessment of intestinal failure and gut absorption | Day -3 and Day 29
  Changes from baseline in bone mineral content by DEXA scan
Assessment of gut regeneration | Day 1 - Day 29
  Measurements of the plasma citrulline (ng/ml)
Plasma Trough concentration (Ctrough) of study drug | Day 1 - Day 29
  Ctrough
Plasma concentration post 72 hours (C72) of study drug | Day 1 - Day 29
  C72

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eliasson J, Hvistendahl MK, Freund N, Bolognani F, Meyer C, Jeppesen PB. Apraglutide, a novel glucagon-like peptide-2 analog, improves fluid absorption in patients with short bowel syndrome intestinal failure: Findings from a placebo-controlled, randomized phase 2 trial. JPEN J Parenter Enteral Nutr. 2022 May;46(4):896-904. doi: 10.1002/jpen.2223. Epub 2021 Sep 7. PMID 34287970